CLINICAL TRIAL: NCT06914375
Title: The Effect of Regular Lentil and Chickpea Intake on Gut Microbiome and Metabolic Health in Healthy Young Adults: A Pilot Randomized Clinical Trial
Brief Title: Effect of Lentils and Chickpeas on Gut Microbiome and Metabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ravi Nagpal, Principal Investigator, Florida State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00005525; 58-3060-4-041 (Other Grant/Funding Number: USDA-ARS)
Record Dates: First submitted 2025-03-30; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Dysbiosis
Keywords: fiber; gut; microbiome; pulses; chickpea; lentil; young adults; transit time; prebiotic; metagenomic; metabolic health
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Chickpea Condition (Experimental): The chickpea (CHK) condition includes a normal diet supplemented weekly with whole-cooked canned chickpeas for 8 weeks (Goya Foods - 120 kcals, 4g fiber, 6g protein per ½ cup). The required intake of chickpeas is determined by stepwise progression of intake according to DGAs 2020-2025 and the participant's gender. Instructions for intake will be provided specifically for each participant and for each week of the study. CHK participants will receive workbooks that contain weekly adherence checklist (dosing diaries), conversion measurements, and copies of RD-prepared recipes outlining various ways to incorporate chickpeas/lentils into their diets each week as meals and/or snacks.
  Interventions: Other: Goya Foods - Canned Chickpeas
- Lentil Condition (Experimental): The lentil condition (LEN) includes a normal diet supplemented weekly with whole-cooked canned chickpeas for 8 weeks (Goya Foods - 80 kcals, 3g fiber, 6g protein per ½ cup). The required intake of chickpeas is determined by stepwise progression of intake according to DGAs 2020-2025 and the participant's gender. Instructions for intake will be provided specifically for each participant and for each week of the study. LEN participants will receive workbooks that contain weekly adherence checklist (dosing diaries), conversion measurements, and copies of RD-prepared recipes outlining various ways to incorporate chickpeas/lentils into their diets each week as meals and/or snacks.
  Interventions: Other: Goya Foods - Canned Lentils
- Control Condition (Active Comparator): The control (CTL) condition will be instructed to consume a normal diet while restricting all pulse intake throughout the study. CTL will receive nutrition education materials in custom workbooks on what pulses are and how to avoid intake.
  Interventions: Other: Control

INTERVENTIONS:
Other: Goya Foods - Canned Chickpeas — Whole-cooked, canned chickpeas supplied by Goya Foods. Provided to participants on a weekly basis in amounts specific to DGAs 2020-2025 and the participant's gender.
  Other Names: chickpeas; CHK
  Arms: Chickpea Condition
Other: Goya Foods - Canned Lentils — Whole-cooked, canned lentils supplied by Goya Foods. Provided to participants on a weekly basis in amounts specific to DGAs 2020-2025 and the participant's gender.
  Other Names: LEN; Lentils
  Arms: Lentil Condition
Other: Control — Participants in the Control condition (CTL) will be asked to consume their standard diet while avoiding any and all pulse intake.
  Other Names: CTL; Control Condition
  Arms: Control Condition

SUMMARY:
The primary goal of this research is to evaluate the effect of daily whole-cooked chickpea and lentil consumption for 8-weeks on gut health, including microbiome-metabolome arrays and gut epithelial/barrier function, in healthy young adults.

Secondary Objectives include:

* To examine the effect of daily whole-cooked chickpea and lentil consumption for 8-weeks on the measures of metabolic health and inflammation in healthy young adults.
* To determine the feasibility of healthy young adults to successfully incorporate and sustain the recommended daily intake of pulses into their diets for eight consecutive weeks

Research Interventions:

Participants will be asked to consume a normal diet supplemented daily with either A) whole-cooked canned lentils, or B) whole-cooked canned chickpeas. The control condition will be instructed to consume a normal diet while restricting all pulse intake throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 30 years old
* Ability to speak and read in English

Exclusion Criteria:

* Intake of antibiotics in the last 3 months
* Intake of pre/pro/postbiotics in the last 3 months
* Current or past (within the last 6 months) user of tobacco, marijuana, or E-cigarette products
* Cardiovascular disease (heart failure, hypertension, hyper/dyslipidemia, past myocardial infarction)
* Gastrointestinal disease (ulcerative colitis, Crohn's disease, diverticulosis, peptic ulcers, small intestinal bacterial overgrowth, fistulas, suspected or known gastric strictures, gastritis, radiation enteritis, GI bleeding, gastric bezoar, recent GI surgery in the last 3 months, etc..),
* Neurological disorders (multiple sclerosis, meningitis, recent stroke) or endocrine disorders (uncontrolled thyroid disorders, growth hormone disorders, adrenal gland disorders, uncontrolled or insulin dependent diabetes - A1C > 9%).
* Food allergy to study foods (pulses or soy, milk, peanuts, tree nuts)
* Regular consumption of pulses (>1 cup/wk for males; >0.5 cup/wk for females)
* Current heavy alcohol use (≥ 15 drinks / week for men, ≥ 8 drinks / week for women)
* Class 3 Obesity (BMI > 40 kg/m2)
* Known to be currently pregnant (self-disclosed).

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Gut Microbiome Diversity | Baseline (day 0) Midpoint (week 4), and endpoint (week 8)
  Collected fecal samples will be used to determine microbiome profiles, including diversity and composition of bacteria.
Change in Oral Microbiome Diversity | Baseline (day 0), endpoint (week 8)
  Collected oral swab samples will be used to determine oral diversity and composition of bacteria in the mouth before and after intervention.
Change in Fecal Metabolome | Baseline (day 0) and Endpoint (week 8)
  The endpoint of fecal metabolomics will be assessed by collecting fecal samples from participants at the beginning and end of the study. These samples will be analyzed using advanced techniques, such as mass spectrometry, to identify and quantify various metabolites present in the feces. The changes in the levels of specific metabolites, which can reflect shifts in gut microbiome composition and metabolic health, will be compared between pre- and post-intervention periods. This analysis will help determine how regular peanut butter intake affects metabolic processes and gut health.
Change in Serum Metabolome | Baseline (day 0), and Endpoint (week 8).
  The endpoint of serum metabolomics will be assessed by collecting blood serum from participants at the beginning and end of the study. These samples will be analyzed using advanced techniques, such as mass spectrometry, to identify and quantify various metabolites present in the serum. The changes in the levels of specific metabolites, which can reflect shifts in gut microbiome composition and metabolic health, will be compared between pre- and post-intervention periods. This analysis will help determine how regular peanut butter intake affects metabolic processes and gut health.

SECONDARY OUTCOMES:
Change in Gut Transit Time | Baseline (day 0), Endpoint (week 8)
  Evaluate changes in gut transit time (measured in minutes) after chickpea, lentil or control conditions from baseline to final analysis, using a blue-dye capsule.
Change in Waist / Hip Circumference | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in waist and hip circumference (centimeters), as well as waist-hip ratio at each study visit before, after and during chickpea, lentil and control conditions.
Change in Lean Mass | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in lean mass (kg). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during experimental (chickpea and lentil) and control conditions.
Change in Habitual Dietary Intake | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Assess changes in habitual dietary intake via 3-day food logs, analyzed using nutrient analysis software (NDSR).
Change in Body Weight | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  The endpoint of body weight (kg) will be measured at each visit to assess changes in weight before, during and after experimental and control conditions.
Change in Lipid Profiles | Baseline (day 0), endpoint (week 8)
  Relevant biomarkers are to be collected via venous blood samples to determine changes in cardiometabolic health including HDL, LDL, total cholesterol, and triglycerides. All will be expressed in units of mg/dL.
Change in Biomarkers of Inflammation | Baseline (day 0), Endpoint (week 8)
  Relevant biomarkers are to be collected via venous blood samples to determine changes in inflammation, including but not limited to C-reactive protein (CRP), IL-1 (Interleukin-1), IL-1 beta, IL-6, IL-10, IL-17, IL-23, Tumor Necrosis Factor Alpha (TNF-a), Interferon-gamma (IFN-Y). All will be expressed in units of pg/mL.
Change in Biomarkers of Intestinal Barrier Function | Baseline (day 0), endpoint (week 8).
  Relevant biomarkers are to be collected via venous blood samples to determine changes in intestinal barrier function including LPS (lipopolysaccharides), LBP (lipopolysaccharide binding protein), CD14, Secretory IgA. All will be expressed in units of pg/mL.
Change in Biomarkers of Appetite | Baseline (day 0), endpoint (week 8)
  Relevant biomarkers are to be collected via venous blood samples to determine changes in appetite including Insulin, Glucagon, glucagon-like peptide 1 (GLP-1), Adiponectin, Leptin, Ghrelin, and Peptide YY. All will be expressed in units of pg/mL.
Change in Rested, Seated Blood Pressure | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  This outcome measure will measure changes in blood pressure taken at rest in the seated position at each visit, before during and after experimental and conrol conditions, expressed as systolic over diastolic blood pressure in units of millimeters of mercury (mmHg).
Change in Fasting Blood Glucose | Baseline (day 0), endpoint (week 8).
  Venous blood samples will be collected to determine changes in fasting blood glucose (expressed as mg/dL).
Dietary Adherence | Daily, baseline through endpoint (week 8)
  Assess adherence to the experimental (chickpeas and lentils) and control condition throughout the study, as determined by dietary adherence logs kept by the participants each week. Adherence is expressed as a daily percent (%) consumption of their assigned condition.
Change in Body Fat Percentage | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including fat mass, expressed as a percentage of total weight (%). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during chickpea, lentil or control conditions.
Change in Total Body Water | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including total body water (TBW) expressed in liters (L). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during chickpea, lentil or control conditions.
Change in Intracellular Fluid | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including intracellular fluid (ICF) expressed in liters (L). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during chickpea, lentil or control conditions.
Change in Extracellular Fluid | Baseline (day 0), midpoint (week 4), endpoint (week 8).
  Evaluate changes in body composition, including extracellular fluid (ECF) expressed in liters (L). This is assessed using a bioimpedance spectroscopy device (ImpediMed SBF7) at each study visit before, after and during chickpea, lentil or control conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Ravinder Nagpal, Ph.D., Principal Investigator — Florida State University
Locations (1):
- Florida State Univresity - The Gut Biome Lab, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Deidentified IPD will not be retain past three years, at the time of this submission the researchers does not plan to make IPD available

REFERENCES:
- See also: The corresponding official Gut Biome Lab website is linked here — https://thegutbiomelab.annescollege.fsu.edu/